CLINICAL TRIAL: NCT05424965
Title: Study to Investigate Signaling Pathways in Placentas of Overweight or Obese Patients and Patients With Gestational Diabetes Mellitus
Brief Title: Cologne Placenta Cohort (CPC)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sarah Appel (Other)
Responsible Party: Sponsor-Investigator, Sarah Appel, Principal Investigator, Universitätsklinikum Köln
Organization: Universitätsklinikum Köln (Other)
Other Study IDs: 14-244
Record Dates: First submitted 2022-01-04; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Obesity, Maternal; Gestational Diabetes Mellitus in Pregnancy
MeSH Terms: conditions — Pregnancy in Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — placenta tissue, maternal blood (plasma, serum, EDTA-blood), umbilical cord blood (plasma, EDTA-blood).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- normal weight without gestational diabetes: BMI < 25; normal glucose tolerance
  Interventions: Other: no intervention
- normal weight with gestational diabetes: BMI < 25; impaired oral glucose tolerance
  Interventions: Other: no intervention
- overweight without gestational diabetes: BMI 25 - 29.9; normal glucose tolerance
  Interventions: Other: no intervention
- overweight with gestational diabetes: BMI 25 - 29.9; impaired glucose tolerance
  Interventions: Other: no intervention
- obese without gestational diabetes: BMI >= 30; normal glucose tolerance
  Interventions: Other: no intervention
- obese with gestational diabetes: BMI >= 30; impaired glucose tolerance
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Aim of the study was to determine if signaling pathways in placentas of mothers affected by overweight/obesity or by gestational diabetes are altered compared to placentas of a control group (normal weight, no gestational diabetes). Moreover, maternal blood and umbilical cord blood were analysed.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* BMI before pregnancy >= 18
* with & without gestational diabetes
* c-section at gestational week 35+0 until 41+6

Exclusion Criteria:

* multiple pregnancy
* maternal serious internal disease
* infections before pregnancy (e.g. HIV, hepatitis B)
* pregnancy-associates diseases (e.g. gestoses, androgen insensitivity syndrome)

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: Obstetrics deptartment of a University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Activity of Wnt signaling pathway in placental tissue | through study completion, about 4 years in total
  Analysis of components of the Wnt signaling pathway; like LRP6 receptor, beta-Catenin, GSK3beta, Wnt ligands (=proteins of interest) and an appropriate protein for normalization.
  Total protein lysates of placental tissue will be used. Analysis will be performed by western blotting and subsequent densitometric analysis. Outcome measure will be [relative protein level of protein or interest/relative protein level of normalization protein].

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Appel, Dr., Principal Investigator — Universitätsklinikum Köln
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No